CLINICAL TRIAL: NCT03598413
Title: A Randomized Controlled Trial of Standard or DHA/EPA Supplemented Enteral Nutrition in Patients Undergoing Laparoscopic Colorectal Surgery
Brief Title: PeRioperative Omega Three and the Effect on ImmuNity
Acronym: PROTEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Daniel White, Surgical Research Fellow, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 18SURN238410
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer; Nutritional Deficiency; Infected Wound; Surgical Site Infection; Complication, Postoperative; Surgery; Surgery--Complications; Sarcopenia; Phagocytic Dysfunction
Keywords: enhanced recovery; perioperative nutrition; macrophages; omega 3 fatty acids
MeSH Terms: conditions — Colorectal Neoplasms; Malnutrition; Wound Infection; Surgical Wound Infection; Postoperative Complications; Sarcopenia; Phagocyte Bactericidal Dysfunction | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Prospective Randomised controlled trial
Who Masked: Investigator
Masking Description: Single blind trial, analysis of all samples blinded to investigation team.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients undergoing standard laparoscopic colorectal resection with no omega-3 enriched peri-operative nutritional support
- Omega-3 (Experimental): Patients in this group will receive 7 days pre and 7 days post surgery of a nutritional supplement enriched with 1.42g/dose of the fish oils EPA and DHA. The supplement is pre-mixed and will be taken twice daily for a total of 14 days.
  Interventions: Dietary Supplement: Omega-3

INTERVENTIONS:
Dietary Supplement: Omega-3 — 200ml, pre-mixed oral nutritional supplement supplying 1.42g per bottle of EPA and DHA.
  Arms: Omega-3

SUMMARY:
Bowel cancer is the second most common cause of cancer-related death in the UK, with 50,000 new cases and over 15,000 deaths annually. Surgery is the mainstay of treatment and the most common complications are an infection of the wound or lungs. These can lengthen hospital stay, reduce the quality of life, and even increase the risk of death. Bowel cancer patients are often malnourished. Optimising nutrition with supplements such as fish-oils can improve the immune response of patients, helping prevent such complications, shorten hospital stay, improve quality of life and overall survival.

DETAILED DESCRIPTION:
Bowel cancer is the second most common cause of cancer-related death in the UK, with 50,000 new cases and over 15,000 deaths annually. Surgery is the mainstay of treatment and the most common complications are an infection of the wound or lungs. These can lengthen hospital stay, reduce the quality of life, and even increase the risk of death. Bowel cancer patients are often malnourished. Optimising nutrition with supplements such as fish-oils can improve the immune response of patients, helping prevent such complications, shorten hospital stay, improve quality of life and overall survival. We are increasingly familiar with the term BMI, body mass index, which we use to categorise obesity in healthcare. A newer term in this realm is that of sarcopenia, a low muscle mass relative to your size, unrelated to your weight or fat density. This can be measured in a number of ways, including on a scan performed routinely in bowel cancer care, a CT scan. Evidence shows that people with low muscle mass, irrespective of their overall weight, experience more complications than those who have healthier amounts of muscle. We hypothesise that patients supplemented with fish oils both before and after surgery will experience an enhancement of their immune response, and subsequently encounter fewer infectious complications, a shorter length of hospital stay and improved quality of life. We also predict fewer patients having extra nutrition before and after surgery will develop sarcopenia and avoid the risks associated with that condition. The trial will only take place in those with bowel cancer who are planned to have a keyhole operation, as this is now the most commonplace approach to surgery. We plan to recruit 40 patients, 20 to receive the supplement, and 20 to form a comparison or control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer undergoing elective laparoscopic colorectal resection.
* Adult aged 18 or over.
* Capacity to consent

Exclusion Criteria:

* Pre-existing diagnosis of Diabetes mellitus, requiring medication.
* Consumption of > 3 alcoholic drinks/day
* Already on omega-3 supplementation
* Pregnant
* Patients on heparin infusion perioperatively
* Patients on immunosuppressive drugs
* Regular / Daily smokers
* Patients requiring a blood transfusion at any point day 7 pre-op to day 1 post operatively.
* Vegan or Vegetarian
* Allergy to cows milk or wheat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Changes in Phagocytosis of pathogens | Baseline [2-4 weeks before surgery], Day of Surgery [day 7 post nutritional supplementation], Day 1 post surgery [day 8 post supplementation].
  Phagocytosis of E.Coli, S.Aureus and Candida measured with flow cytometry
Changes in cell membrane composition | Baseline [2-4 weeks before surgery], Day of Surgery [day 7 post nutritional supplementation], Day 1 post surgery [day 8 post supplementation].
  Using gas chromatography, measuring the percentage of omega-3 within cell membranes

SECONDARY OUTCOMES:
Infectious complications | 30 days
  Descriptions laid out in supplement 1 for diagnostic criteria
Non-infectious complications | 30 days
  Descriptions laid out in supplement 1 for diagnostic criteria
Length of hospital stay | A maximum of 90 days
  Length of stay in days as per electronic discharge records
Sarcopenia | Baseline [Pre-operative staging CT scan] and 6 month +/-2 months
  Changes in body composition measured on CT scan
Quality of Life (EORTC: QLQC30) | Baseline and 3 weeks post surgery +/- 7 days
  Quality of life questionnaire EORTC: QLQC30. A 30 element validated questionnaire. Symptoms are grouped into scales: Physical Function, Role Function, Emotional Function, Cognitive Function, and Social Function. In addition symptom scales including: Fatigue, Nausea, vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea, and financial difficulties. 28 of the scales range from 1 to 4, 4 being most symptomatic, 1 least so. The 2 remaining scales for overall health and quality of life are scaled 1-7, with 7 being the best and 1 the worst. The 30 questions can be combined for a global score, in which instance the 2 global scales are reversed so that 7 becomes the worst quality of life or health and 1 the best.
Changes in Hand grip strength | Baseline [Pre-operative staging CT scan] and 6 month +/-2 months
  Physical measurement of hand grip strength using hand dyanamometer to assist in diagnosis of sarcopenia / functional status.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Ethical approval allows for sharing of anonymised data with collaborators at the University of Surrey.